CLINICAL TRIAL: NCT04937556
Title: Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effect of the Lactobacillus Probiotic Strain in the Immune Response in Participants Positive for SARS-CoV-2 (Severe Acute Respiratory Syndrome-Coronavirus-2) Infection.
Brief Title: Evaluation of a Probiotic Supplementation in the Immune Response of Participants With COVID-19 (Coronavirus Disease).
Acronym: PROVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ProbiSearch SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COV/21.02
Record Dates: First submitted 2021-06-14; First posted 2021-06-24 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Zinc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic: Lactobacillus salivarius + Vit D + Zinc (Active Comparator): Lactobacillus strain during 28 days, approximately 1*10E9 colony forming unit (CFU) of L. salivarius in 1 capsule per day.
  Interventions: Dietary Supplement: Probiotic: Lactobacillus salivarius + Vit D + Zinc
- Placebo (Placebo Comparator): Placebo supplement in 1 capsule per day during 28 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic: Lactobacillus salivarius + Vit D + Zinc — A mixture of 1*10E9 colony forming unit (CFU) of Lactobacillus salivarius + Vit D + Zinc citrate in 1 capsule will be daily administrated during 28 days.
  Arms: Probiotic: Lactobacillus salivarius + Vit D + Zinc
Dietary Supplement: Placebo — Placebo in 1 capsule will be daily administrated during 28 days.
  Arms: Placebo

SUMMARY:
An interventional, randomized, double-blind, placebo-controlled study will be conducted to investigate the effect of a probiotic strain on the immune response in participants positive for SARS-CoV-2 infection.

The study duration will be 28 days, which includes 4 weeks product administration. Participants will be randomized assigned to one of the two study groups: the control group with placebo consumption and a probiotic consumption group.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18-65 years).
* Mild infection by SARS-CoV-2 detected by PCR or Antigen.
* Onset of COVID-19 symptoms up to 5 days before the day of inclusion
* Without hospitalization or oxygen supplementation on the day of inclusion.
* Signed written informed consent

Exclusion Criteria:

* Serious SARS-CoV-2 infection requiring hospitalization or oxygen supply
* Chronic diseases under regular medication (eg asthma, allergic rhinitis ...)
* Congenital or acquired immunodeficiency
* Body Mass Index (BMI)> 30
* Coagulation disorders
* Short bowel syndrome or any surgery on the gastrointestinal tract.
* Metabolic disorders (diabetes, etc.).
* Heart failure and cardiac medical history
* Pregnant women.
* HIV positive.
* Immunocompromised
* History of significant gastrointestinal diseases
* Use of other probiotics during the last month.
* Uncertainty about the willingness or ability of the participant to comply with the requirements of the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Concentration of specific IgM (Immunoglobulin M) and IgG (Immunoglobulin G) antibodies for the SARS-CoV-2 virus. | 1 month

SECONDARY OUTCOMES:
Levels (pg/ml) of pro-inflammatory and anti-inflammatory markers in blood serum. | 1 month
Duration of the symptoms produced by the SARS-CoV-2 infection | 1 month
Severity of symptoms produced during SARS-CoV-2 infection | 1 month
  Severity of symtoms will be analysed for fever (Tª>38ºC) and gastrointestinal symptons (Bristol scale).
Percentage of participants with a negative result in the SARS-CoV-2 detection test by PCR (Polymerase Chain Reaction) at visit 2 | 1 month
Percentage of participants with worsening of lower respiratory tract infections | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Infanta Leonor, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.probisearch.com